CLINICAL TRIAL: NCT06723210
Title: Parkinson´s Disease: Correlation Analysis Between the Cardinal Motor Symptoms of the Illness and the Male Patients´ Body Composition
Brief Title: Parkinson and the Males Body Composition
Acronym: PD&MBC
Status: Completed | Type: Observational
Sponsor: University of Oviedo (Other)
Collaborators: University of Leon (Unknown)
Responsible Party: Principal Investigator, Luis Santos, PhD, University of Oviedo
Other Study IDs: ETICA-ULE-081-2024
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Neurodegenerative Disease
Keywords: Movement Disorders; Components of the Human Body
MeSH Terms: conditions — Neurodegenerative Diseases; Movement Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: The patients were assigned to the same group because the study´s design only demands to create one group of patients.

SUMMARY:
The main aim of the present study was to ascertain the type of relationship (dependency or independency) among some of the cardinal motor symptoms of the Parkinson´s disease (PD) and the body composition (BC) variables of a group of the male PD´s patients, using the bioelectrical impedance analysis.

ELIGIBILITY:
Inclusion Criteria:

(I) Males with diagnosis of idiopathic PD and rated 1-3 on the Hoehn and Yahr Scale.

(II) No type of dementia as assessed by the mini-mental state examination. (III) Between 50 and 69 years old (a specific range of ages of the illness´s onset).

(IV) Between one and five years diagnosed with the illness. (V) Able to stand for two min without assistance. (VI) Able to walk teen m without assistance.

Exclusion Criteria:

(I) Do not meet the eligibility criteria. (II) Suffer a neurological disease other than Parkinson´s disease.

Ages: 50 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is focused on the Parkinson´s disease male patients
Study Population: A group of fifteen male patients with idiopathic Parkinson´s disease participated in the project.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
The body composition variables or the bioelectrical impedance variables | From February 2025 to February 2025
  weight (kg), fat-free mass in absolute terms (FFMa) (kg), fat-free mass in relative terms (FFMr) (normalized per kg of body mass -kg/kg of body weight-), fat-free mass of the right arm (FFMRA) (kg), fat-free mass of the left arm (FFMLA) (kfg), difference between the FFMRA and the FFMLA (%), fat-free mass of the right leg (FFMRL) (kg), fat-free of the mass left leg (FFMLL) (kg), difference between the FFMRL and the FFMLL (%), body fat mass (BFM) (kg), skeletal muscle mass (SMM) (kg), body mass index (BMI) (kg/m2), percentage body fat (PBF) (%), total body water in absolute terms (TBWa) (L), total body water in relative terms (TBWr) (normalized per kg of body mass -kg/kg of body weight-), total water of the right arm (TWRA) (L), total water of the left arm (TWLA) (L), difference between the TWRA and the TWLA (%), total water of the right leg (TWRL) (L), total water of the left leg (TWLL) (L), difference between the TWRL and the TWLL (%), intracellular water (ICW) (L), extracellular
The Movement Disorder Society-Unified Parkinson´s Disease Rating Scale (MDS-UPDRS)) | From February 2025 to February 2025
  MDS-UPDRS: Spanish validated version of the MDS-UPDRS. The possible score ranges from 0 to 72 points whereby 0 points represent a healthy status and the more points, the worse health status.
The Ten-Meter Walk Test | From February 2025 to February 2025
  The Ten-Meter Walk Test: performance measure used to assess walking speed in meters per second over a short distance (10 meters).
Step length | From February 2025 to February 2025
  The step length of the patients will be determined using kinematic gait analysis during the TMWT, utilizing the OptoGait system (Microgait, Optogait, v.1.12.21, Italy). The step length of the patients will be determined in cm. This system consists of transmitter and receiver bars equipped with optical sensors operating at a frequency of 1000 Hz, which will be positioned along the ten-meter walking corridor, from meter two to meter seven.
: Spanish validated version of the Disability of the Arm, Shoulder and Hand (DASH) | From February 2025 to February 2025
  DASH: Spanish validated version of the Disability of the Arm, Shoulder and Hand. The possible score ranges from 0 (which means no disability) to 100 (which means most severe disability). Higher scores indicate a greater level of disability and severity, whereas, lower scores indicate a lower level of disability.
The Timed up and Go Test (TUG) | From February 2025 to February 2025
  TUG: The TUG measures of functional mobility that was initially developed to identify mobility and balance impairments. Participants takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees, as fast as they can (the time of the test is determined in sec).
Handgrip Strength of both hands. | From February 2025 to February 2025
  Handgrip Strength of both hands: manual dynamometer measured in kilograms.
Static posturography | From February 2025 to February 2025
  Static posturography, assessed by measurement of the center of pressure (CoP). These CoP parameters; Length, in mm, Area in mm2 and Speed, Xspeed and Yspeed in m/s will be combined to report the patient´s static posturography.
The nine holes peg test (9-HPT) | From February 2025 to February 2025
  The nine holes peg test (9-HPT) is a brief, standardized, quantitative test of upper extremity function. Both the dominant and non-dominant hands are tested twice. The patient is seated at a table with a small, shallow container holding nine pegs and a wood or plastic block containing nine empty holes. On a start command when a stopwatch is started, the patient picks up the nine pegs one at a time as quickly as possible, puts them in the nine holes, and, once they are in the holes, removes them again as quickly as possible one at a time, replacing them into the shallow container. The total time to complete the task is recorded in minutes. Two consecutive trials with the dominant hand are immediately followed by two consecutive trials with the non-dominant hand. The score for the 9-HPT is an average of the four trials. The two trials for each hand are averaged, converted to the reciprocals of the mean times for each hand and then the two reciprocals are averaged.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oviedo, Oviedo, Spain, Spain